CLINICAL TRIAL: NCT00302549
Title: To Compare the Efficacy and Safety of FK506 vs IVC in the Treatment of Class
Brief Title: To Compare the Efficacy and Safety of FK506 vs IVC in the Treatment of Class III-IV LN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0602
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2008-07

CONDITIONS: Lupus Nephritis
Keywords: Tacrolimus; Cyclophosphamide; Treatment; Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FK506 (Active Comparator)
  Interventions: Drug: FK506

INTERVENTIONS:
Drug: FK506 — FK506,0.1mg/kg/d
  Other Names: Tacrolimus,Prograf

SUMMARY:
1. To compare the efficacy of FK506 vs intravenous cyclophosphamide pulses in the treatment of class III-IV LN.
2. To compare the safety and tolerability of FK506 vs intravenous cyclophosphamide pulses in the treatment of class III-IV LN.
3. To explore the dosing of FK506 and its effective range of blood concentration.

DETAILED DESCRIPTION:
Corticosteroid combined with cytotoxic drugs has been regarded as the conventional therapy for Class IV Lupus Nephritis (LN), because of its efficacy in improving patients' long term survival. However, this treatment fails in some patients, especially those who present with significant vascular lesion. In addition, cyclophosphamide (CTX) has severe side effects with a high incidence of marrow inhibition and infection.FK506 (Tacrolimus) is a new calcineurin inhibitor. Similar to Cyclosporine (CsA), it inhibits the production of IL-2 and activation of T cells. Furthermore, it has an added value of inhibiting the production of IL-10 from Th2 cells, thus reducing the production of auto antibodies from B cells.It also exerts its specific immunosuppressive effects through CsA-insensitive pathway. FK506 could inhibit not only the activation of naive T cells but also the activation and proliferation of primed T cells.FK506 is 10 -100 times more powerful than CsA in inhibiting the activation of T cells.Animal studies on MRL/lpr mice LN model demonstrated that FK506 could significantly depress the excretion of urine protein and the level of serum anti-dsDNA, inhibit glomerular cellular proliferation and formation of crescents, and reduce the deposits of immune complex.

A preliminary study showed that FK506 was significantly effective on patients with IV LN,as indicated by rapid reduction of urine protein, increase in serum albumin, decrease in auto antibodies together with remission of lesion activity of the renal tissue. However, the drawbacks of this study were the small sample size and the lack of a controlled group. Hence, a multi-center controlled study comparing FK506 with cytotoxic agents to evaluate the efficacy and safety of FK506 on patients with III or IV LN, and explore the effective range of FK506 blood concentration and the appropriate target patient population would be needed.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with a diagnosis of Systemic Lupus Erythematosus (SLE) according to the criteria of American Rheumatic Association, 1982 (Appendix 1) aged between 18-65 years, and whose score of SLE-DAI (Disease Active Index, Appendix 2) is greater than 10.
2. Patients diagnosed to have class III or IV LN by renal biopsy, according to the WHO classification criteria (1995, Appendix 3) within 3 month and have significant active pathological lesion.
3. Patients with a proteinuria ≥ 2g/24h, and an active urine sediment (Hematuria with white cells and casts in urine).
4. Patients who signed written informed consent form (patients less than 18 years old with their parents/legal representative's signatures), and have given their consent to follow all study procedures and follow-up.

Exclusion Criteria:

1. Patients who have received treatment of cytotoxic drugs such as CTX, Mycophenolate mofetil (MMF) cyclosporine for more than 1 week within three months, but Azathioprine (AZa) are accepted.
2. Patients with serum creatinine > 3 mg/dl（265μmol/L）.
3. Patients with severe infection or central nervous system symptoms.
4. Patients who have impaired liver function, with ALT/GPT or AST/GOT twice more than the normal upper limit or who have active hepatitis.
5. Patients who have abnormal glucose, with a fasted blood glucose > 6.2 mmol/L or post meal blood glucose > 11.2 mmol/L.
6. Patients who are pregnant or lactating.
7. Patients who are known to be allergic to a macrolide.
8. Patients who use Erythromycin, Fluconazole, Ethinylestradiol, Rifampicin, and Carbamazepine.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2004-05; Primary Completion 2005-05 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of FK506 vs intravenous cyclophosphamide pulses in the treatment of class III-IV LN | 6 months

SECONDARY OUTCOMES:
To compare the safety and tolerability of FK506 vs intravenous cyclophosphamide pulses in the treatment of class III-IV LN and to explore the dosing of FK506 and its effective range of blood concentration. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lei-shi Li, M.D., Study Director — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China